CLINICAL TRIAL: NCT00000929
Title: Phase I Rectal Microbicide Study
Brief Title: A Study of the Effects of Advantage 24 on the Rectum
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Prevention
Other Study IDs: HIVNET 008; 11715 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Sexual Partners; Homosexuality, Male; Anti-Infective Agents; Patient Compliance; Nonoxynol; Rectum
MeSH Terms: conditions — HIV Infections; Homosexuality, Male; Patient Compliance | interventions — Nonoxynol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Nonoxynol-9

SUMMARY:
The purpose of this study is to see if it is safe and acceptable for homosexual male couples, where both partners have the same HIV status, to use Advantage 24 during anal intercourse. Advantage 24 is a spermicide (a chemical that kills sperm).

Much research and development is being done with chemicals that can be controlled by the receptive partner to prevent the spread of HIV and other sexually transmitted diseases (STDs). Advantage 24 currently is used in the vagina as a form of birth control. The safety of Advantage 24 is particularly important for HIV-positive men because they have a greater chance of serious reaction to Advantage 24 due to other HIV-related conditions.

DETAILED DESCRIPTION:
Chemical barriers which can be controlled by the receptive partner to prevent transmission of HIV and other sexually transmitted diseases (STDs) are among the highest priorities for research and development. Advantage 24 is a contraceptive gel containing nonoxynol-9 (N-9). This study provides information on the safety of N-9 in a bioadhesive gel formulated for use by MSM during anal intercourse. Safety is assessed for both HIV-positive and HIV-negative men because HIV-positive men may be at increased risk for toxicity due to other HIV-related conditions.

Participants are divided into 4 cohorts depending on their serostatus and whether they are the insertive or receptive partner. Participants apply Advantage 24 once or twice a day for 5 weeks and 4 times a day for the sixth week. Check-in visits, which include a genital exam, are performed at Weeks 1, 2, 4, 5, and 7. More complete physical evaluations, including anoscopy for receptive partners and blood tests, are performed at Weeks 3, 6, and 8.

ELIGIBILITY:
Exclusion Criteria

Co-existing Condition:

Participants with the following symptoms or conditions are excluded:

* Positive HSV-2 serology (HIV-negative participants only).
* Positive syphilis by Venereal Disease Research Laboratory (VDRL) serology and Fluorescent Treponemal Antibody (FTA) or Microhemagglutination Assay (MHA).

Receptive partners with the following additional symptoms or conditions are excluded:

* Rectal gonorrhea or chlamydia by culture.
* Active rectal inflammation, ulceration, or fissures.

Insertive partners with the following additional symptoms or conditions are excluded:

* Penile or urethral irritation, rashes, or lesions.
* Penile or scrotal piercing.

Concurrent Medication:

Excluded for receptive partners:

-

Anticoagulant, including warfarin and heparin.

Participants with the following prior conditions are excluded:

* Sensitivity or irritative symptoms when using N-9 or when exposed to latex.
* Three or more Herpes Simplex 2 Virus (HSV-2) outbreaks within 12 months prior to screening (HIV-positive participants only).
* One or more HSV-2 outbreaks within 6 months prior to screening (HIV-positive participants only).

Receptive partners with the following additional prior conditions are excluded:

* Diagnosed inflammatory bowel disease, ulcerative colitis, Crohn's disease, or rectal malignancy.
* Diagnosed bleeding disorder, including hemophilia and thrombocytopenia.
* Rectal surgery including fistulectomy.
* Prosthetic heart valve or diagnosis of a valvular abnormality.
* Hemorrhoidectomy within 6 months prior to screening.
* Rectal burning, tenesmus, bleeding, or irritation in the week prior to screening.
* Diarrhea (more than 3 stools per day) in the week prior to screening.
* Use of rectally-inserted sex toys, practiced receptive fisting, or rectal douching in the week prior to screening.

Insertive partners with the following additional prior conditions are excluded:

Urethral burning or discharge in the week prior to screening.

Prior Medication:

Excluded for receptive partners:

Use of laxatives in the week prior to screening.

Participants meet the following criteria:

* HIV-negative or HIV-positive; participant's partner must be the same serostatus.
* Plan to have anal intercourse only with the study partner for the duration of the study. During all episodes in which Advantage 24 is used, one partner is exclusively insertive and the other partner is exclusively receptive.
* Sexual partner of at least 3 months is eligible and agrees to participate.
* Agree to use non-N-9 lubricant and condoms for all episodes of anal intercourse.
* Avoid use of Advantage 24 for purposes other than specified by the protocol.

Receptive partners meet the following additional criteria:

* Plan to have receptive anal intercourse with the study partner with Advantage 24 applied rectally, and using N-9 lubricant and condoms, at the couple's usual frequency (at least 3 times per week).
* Agree to apply the specified amount of Advantage 24 daily to the rectum.
* Avoid use of laxatives, use of rectally-inserted sex toys, receptive fisting, and rectal douching.

Insertive partners meet the following additional criteria:

* Plan to have insertive anal intercourse with the study partner with Advantage 24 applied to the glans of the penis, and using non-N-9 lubricant and condoms, at the couple's usual frequency (at least 3 times per week).
* Agree to apply the specified amount of Advantage 24 daily to the penis.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70
Dates: Study Completion 1999-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Connie Celum, Study Chair; Susan Buchbinder, Study Chair
Locations (1):
- Univ of Washington, Seattle, Washington, United States